CLINICAL TRIAL: NCT06348342
Title: The Effectiveness of Pelvic Floor Muscle Exercises and Core Exercises in Menopausal Women With Stress Urinary Incontinence
Brief Title: Pelvic Floor Muscle Exercises and Core Exercises in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assist. Prof, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TÜTF-GOBAEK 2023/24
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Stress Urinary Incontinence; Kegel Exercises; Core Strength
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Before starting the research, four groups of mothers will be randomly formed. As a randomization method, mothers who meet the sampling inclusion criteria determined in the research will be identified and listed. Individuals to be taken into two groups will be determined by randomization method from the random numbers table. (http://www.stattrek.com/statistics/randomnumbergenerator.aspx).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention)
- Kegel (Experimental): Kegel exercises
  Interventions: Other: Pelvic Floor Muscle Exercise
- Core (Experimental): Core exercises
  Interventions: Other: Core Exercise
- Kegel+core (Experimental): Kegel and core exercises
  Interventions: Other: Pelvic Floor Muscle Exercise; Other: Core Exercise

INTERVENTIONS:
Other: Pelvic Floor Muscle Exercise — Training for PFME will be given orally and will cover the importance of FME and how to do the exercises, as well as the conditions and frequency of doing the exercises. You will be told that the exercise should be done when the bladder is empty, three times a day (morning, noon and evening) and repeated 10 times in each set. In the first week of exercise, the pelvic floor muscles will be contracted for 3 seconds and relaxed for 3 seconds, and will be increased by 1 second each week. It will be explained that from the 8th week onwards, it will be done by contracting for 10 seconds and relaxing for 10 seconds and will continue. It will be stated that the learning process of pelvic floor muscle exercise may take 6 weeks to 6 months. It will be stated that this exercise should be applied throughout their lives for the sustainability of PFM strength. The training is planned to last approximately 20 minutes. PFME will last for two months. Women in menopause will be given an exercise chart.
  Arms: Kegel; Kegel+core
Other: Core Exercise — Activating the contraction of the deep core muscles TrA and mutifidus without disrupting breathing forms the basis of core stabilization exercises. To teach the "abdominal hallowing" maneuver, which enables the activation of these muscles, patients will be shown a picture of the TrA muscle and asked to contract their lower abdominal muscles while lying on their back in the hook position. During the maneuver, care will be taken to ensure that no movement occurs in the trunk and pelvis and that diaphragmatic breathing continues. After the abdominal hallowing maneuver is taught, the exercises will be progressed gradually. A home exercise program will be given for this. The 7-level exercise program recommended by Hagins et al. will be used as a home exercise program. The movements in this program load more moments on the muscles that stabilize the lumbar spine as the levels progress. The stages of the exercise program are shared in the brochure to be given to the patients.
  Arms: Core; Kegel+core

SUMMARY:
The prospective and four-arm randomized controlled study was conducted on n = 136 (34 = control, 34 = kegel, 34 = core, 34 = kegel+ core group) menopausal women at Trakya University Health Research and Application Center Urology Polyclinic between Oct 2023 and June 2024. In the first interview, the researcher will apply an information form to all four groups, asking about personal information, habits, bladder irritants and fluid intake-related features, obstetric, gynecological and systemic disease-related features, and stress urinary incontinence-related features. This form will only be filled at the beginning. In addition, the "Pelvic Floor Distress Scale (PFDI)" and "Pelvic Floor Impact Questionnaire (PFIQ)" will be applied and will be repeated by the executive researcher at the 1st, 2nd and 3rd controls. It will be terminated at the 3rd follow-up. Descriptive statistics, Pearson, Spearman's correlation, and regression analyzes will be used in the analysis of research data.

DETAILED DESCRIPTION:
In this prospective, randomized-controlled study, menopausal women over the age of 45 who applied to Trakya University Health Research and Application Center Urology Polyclinic with complaints of stress urinary incontinence (stage 1-2) and who do not require surgical or medical treatment of stress urinary incontinence were included in the case and intervention groups. will be divided into four groups:

In the first interview, the researcher will apply an information form to all four groups, asking about personal information, habits, bladder irritants and fluid intake-related features, obstetric, gynecological and systemic disease-related features, and stress urinary incontinence-related features. This form will only be filled at the beginning. In addition, the Pelvic Floor Distress Scale (PFDI); and Pelvic Floor Impact Questionnaire (PFIQ); will be applied and will be repeated by the executive researcher at the 1st, 2nd and 3rd controls. It will be terminated at the 3rd follow-up.

All four groups will be given a 3-day voiding diary, which will be requested at the check-up and must be filled out at home for 3 consecutive days (a voiding diary will be given at each follow-up and they will be asked to bring it at the 1st, 2nd and 3rd follow-up a month later) and will be monitored by the leading researcher. It will be terminated at the 3rd follow-up.

At the 3rd follow-up, where the study was terminated; Trakya University Faculty of Medicine Urology Department, which will perform routine control examinations of diagnosed patients and is involved in the study. Faculty Member Assoc. Dr. Hakan AKDERE and Op. Dr. Hakan ÇAKICI at Private Optimed Hospital Urology Department. Urogynecological evaluation tests (stress test, uroflowmetry, pelvic floor muscle strength measurement, digital palpation) will be requested and will be performed by the researchers in the examination room of the Urology Polyclinic of the applied hospital, paying attention to the privacy of women. The requested urogynecological evaluations will be requested in the 3rd follow-up and are the tests included in the patient follow-up protocol of the specified diagnosis. No evaluation test other than routine evaluation tests is specified.

Pelvic Floor Muscle Exercise (PFME/ Kegel Exercise): Training for PFME will be given orally and will cover the importance of PFME and how to do the exercises, as well as the conditions and frequency of doing the exercises. You will be told that the exercise should be done when the bladder is empty, three times a day (morning, noon and evening) and repeated 10 times in each set. In the first week of exercise, the PFM will be contracted for 3 seconds and relaxed for 3 seconds, and will be increased by 1 second each week. It will be explained that from the 8th week onwards, it will be done by contracting for 10 seconds and relaxing for 10 seconds and will continue. It will be stated that the learning process of pelvic floor muscle exercise may take 6 weeks to 6 months. It will be stated that this exercise should be applied throughout their lives for the sustainability of PFM strength. The training is planned to last approximately 20 minutes. PFME will last for two months. Women in menopause will be given an exercise chart (about how many times a day they should exercise) to guide them in their exercise activities at home.

Core Exercise: Activating the contraction of the deep core muscles TrA and mutifidus without disrupting breathing forms the basis of core stabilization exercises. To teach the abdominal hallowing; maneuver, which enables the activation of these muscles, patients will be shown a picture of the TrA muscle and asked to contract their lower abdominal muscles while lying on their back in the hook position. During the maneuver, care will be taken to ensure that no movement occurs in the trunk and pelvis and that diaphragmatic breathing continues. After the abdominal hallowing maneuver is taught, the exercises will be progressed gradually. A home exercise program will be given for this. The 7-level exercise program recommended by Hagins et al. will be used as a home exercise program. The movements in this program load more moments on the muscles that stabilize the lumbar spine as the levels progress. The stages of the exercise program are shared in the brochure to be given to the patients. The aim of the exercise program is to complete the movements without disrupting the abdominal hallowing. Each patient, whose urogynecological values are completed and who meets the diagnosed criteria, will visit the physiotherapist researcher at the Department of Physical Therapy and Rehabilitation, Faculty of Health Sciences, after Trakya University Health Practice and Research Hospital, to teach the abdominal hallowing maneuver and to determine at what level they will start stabilization exercises. Patients will be given a program of 3 movements, one level below and one above the level they can achieve. The program, which will last 15 minutes in total, with each movement being five minutes, will be done 3 days a week, and the core exercise will last for two months. Patients will be evaluated by a physiotherapist once a month to evaluate the activation of the TrA muscle and their exercise programs will be updated.

In the stress test, if the bladder is full and there is a feeling of urination, the patient will first be evaluated in the lithotomy position on the examination table, and the same procedure will be performed while standing, by asking for strong straining and coughing, by increasing the intra-abdominal pressure, and visually visualizing whether there is urine leakage.

After the stress test; With the uroflowmetry evaluation test, the woman will be seated on the upper toilet, under which the uroflowmetric device is located, and the researcher will be asked to urinate completely with the start. After urinating completely, the process will be terminated with the finish from the researcher. With this method, urination volume, flow duration, maximum flow rate, time to reach maximum speed, average flow rate and urination time values will be measured and the values will be taken through the software to which the device is connected.

Pelvic Floor Muscle Strength Measurement: With the device called perinometry, which measures the pelvic floor muscle strength, the vaginal probe, which belongs only to the woman, will be placed 3 cm inside the chamber, and the pelvic floor muscle strength will be evaluated by giving the woman a muscle command to the pelvic floor muscles.

Digital Palpation is a subjective method applied by vaginal touch that evaluates the strength and endurance (maximum duration of contractions) of the pelvic floor muscles. Evaluation by digital palpation will be performed using the Modified Oxford Classification.

Evaluation of PTK strength by digital examination (Modified Oxford scoring) PTK strength Muscle strength 0: No contraction Muscle strength 1: Contraction is minimal, able to hold fingers for less than 1 second.

Muscle strength 2: Contraction is weak, there is no elevation of the fingers and can hold for 1-3 seconds.

Muscle strength 3: With contraction, the doctor's fingers are lifted up to the posteriorvaginal wall, can hold for 4-6 seconds, can repeat 3 times.

Muscle strength 4: The doctor's fingers rise up to the posterior vaginal wall, there is a feeling of more intense pressure on the fingers and can hold it for 7-9 seconds, repeating it 3 times.

Muscle strength 5: Can make one strong contraction lasting 10 seconds and repeat 4 or more times.

The type of stress incontinence will be determined after the evaluation tests applied during the initial interview. Urogynecological evaluation tests and Pelvic Floor Distress Scale (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ) will be repeated at the 1st, 2nd and 3rd controls. Initially, randomly assigned intervention groups will be given exercises that strengthen the pelvic floor muscles (kegel exercise - applied) and core exercise training (applied) after urogynecological evaluation tests, according to the exercise type of the groups. Initially, all randomly assigned groups will be instructed to come for a check-up once a month for 3 months after the urogynecological evaluation tests.

The control group will not do kegel or core exercises and routine treatment processes will continue. Intervention 1 (kegel exercise group only) will only be given exercise training that strengthens the pelvic floor muscles (kegel exercise - applied). Intervention 2 (group doing only core exercise) will be given exercise training that strengthens only the abdominal muscles (core exercise - applied). Intervention 3 (kegel exercise and core exercise group) will be given exercise training (kegel exercise and core exercise - applied) that strengthens the pelvic floor muscles and abdominal muscles.

An exercise tracking chart will be given to all four groups. The follow-up chart will be filled out group-specific (intervention 1: kegel, intervention 2: abdomen and intervention 3: kegel + abdomen) every day, 3 times a day for 3 months, and will be delivered to the researchers at each follow-up, giving detailed information about the form. The 1st, 2nd and 3rd follow-ups after the beginning will be completed with one month intervals for a total of 2 months of follow-up, and the recovery status after exercise treatment will be evaluated with urogynecological evaluation tests. Participants will be followed up by phone once a week for control purposes.

Survey Form: Data collection form prepared by the researcher by scanning the literature; It consists of a total of 55 questions to determine the patients' socio-demographic characteristics, habits, characteristics regarding bladder irritants and fluid intake, characteristics regarding obstetric-gynecological and systemic disease history, and characteristics regarding stress urinary incontinence.

Pelvic Floor Distress Inventory (PFDI - Pelvic Floor Distress Inventionary): PFDI is a symptom questionnaire consisting of 20 items used to measure the degree of discomfort caused by pelvic symptoms in women. Each item consists of 4 options (Not at all, Rarely, Moderately, Quite a lot) and is given a score between 1 and 4. PFDI consists of 3 subscales.

* POPDI-6 (Pelvic organ prolapse distress inventory): It consists of 6 questions and the presence and degree of pelvic organ prolapse symptoms are questioned.
* UDI-6 (Urinary distress inventory): In this sub-dimension, urinary stress incontinence, detrusor overactivity and extra-bladder obstructions are questioned. In addition, according to patients UDI scores; Those with a UDI1 score>1 are classified as having frequency urinary incontinence, those with a UDI2 score>1 as having urge urinary incontinence, those with a UDI3 score>1 as having stress urinary incontinence, those with a UDI2+UDI3 score>2 as having mixed urinary incontinence, and those with a UDI5 score>1 as having urinary retention. .
* CRADI-8 (Colo-rectal-anal distress inventory): It consists of 8 questions asking about symptoms such as constipation, fecal incontinence and flatus incontinence. The average scores of the items in each subscale are calculated, these scores are multiplied by 25, and PFDI subscale scores ranging from 0 to 100 are calculated. Then, the 3 subscale scores are summed to obtain the PFDI total score, which ranges from 0 to 300. A higher score indicates poorer health status.

Pelvic Floor Impact Questionnaire (PFIQ Pelvic Floor Impact Questionnaire): PFIQ is a pelvic floor quality of life questionnaire used to evaluate the effects of bowel, bladder and/or pelvic symptoms on the individual's daily living activities, social relationships and emotions. Each item consists of 4 options (Not at all, Rarely, Moderately, Quite a lot) and is given a score between 0 and 3. The PFIQ scale also consists of 3 subscales.

* POPIQ-7 (Pelvic organ prolapse impact questionnaire): In this subscale consisting of 7 questions, it is questioned how pelvic organ prolapse affects the patient during travel, social activity and physical activity and the impact of this situation on emotional health.
* IIQ-7 (Incoinence impact questionnaire): In this subscale consisting of 7 questions, it is questioned how urinary incontinence during travel, social activity and physical activity affects the patient and the impact of this situation on his emotional health.
* CRAIQ-7 (Colo-rectal-anal impact questionnaire): In this sub-dimension, consisting of 7 questions, it is questioned how bowel complaints affect the patient during travel, social activity and physical activity, and the impact of this situation on emotional health.

The average scores of the items in each subscale are calculated and these scores are multiplied by (100/3) and PFIQ subscale scores ranging from 0 to 100 are calculated. Then, the 3 subscale scores are summed to obtain the PFIQ total score, which ranges from 0 to 300. A higher score indicates poorer health status.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study,
* Those over the age of 45 who are in menopause,
* Women with coitus (+),
* Body mass index < 30 kg/m2,
* Not addicted to alcohol or drugs,
* Experiences recorded unintentional leakage more than once a week,
* Those diagnosed with Stage I-II stress urinary incontinence complaints, Patients whose stress incontinence does not require surgical or medical treatment will be included in the study.

Exclusion Criteria:

* Those who do not volunteer to participate in the study,
* Women who are under the age of 45 and are not in menopause,
* Women with (-) coitus,
* Having a pacemaker installed,
* Presence of a device implanted in the pelvis or hip joint(s),
* Having had pelvic or abdominal surgery in the last 6 months,
* Having a neurological or psychiatric disease,
* Having a urinary tract infection,
* Body mass index >30 kg/m2,
* Those who are addicted to alcohol or drugs,
* Not experiencing any recorded unintentional leakage events more than once a week,
* Those diagnosed with Stage III-IV Stress urinary incontinence complaints,
* Patients requiring surgical and medical treatment of stress incontinence will not be included in the study.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is gender-focused because it is carried out specifically for the menopause period.
Enrollment: 136 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pelvic floor evaluated using the Pelvic Floor Distress Inventory (PFDI - Pelvic Floor Distress Inventionary) | change from baseline and 1, 2, and 3 months of practice
  PFDI is a symptom questionnaire consisting of 20 items used to measure the degree of discomfort caused by pelvic symptoms in women. Each item consists of 4 options (Not at all, Rarely, Moderately, Quite a lot) and is given a score between 1 and 4. PFDI consists of 3 subscales.
Pelvic floor impact evaluated using the Pelvic Floor Impact Questionnaire (PFIQ Pelvic Floor Impact Questionnaire) | change from baseline and 1, 2, and 3 months of practice
  PFIQ is a pelvic floor quality of life questionnaire used to evaluate the effects of bowel, bladder and/or pelvic symptoms on the individual's daily living activities, social relationships and emotions. Each item consists of 4 options (Not at all, Rarely, Moderately, Quite a lot) and is given a score between 0 and 3. The PFIQ scale also consists of 3 subscales.

SECONDARY OUTCOMES:
Urinary incontinence evaluated using the Stress Test | change from baseline and 1, 2, and 3 months of practice
  the bladder is full and there is a feeling of urination, the patient will first be evaluated in the lithotomy position on the examination table, and the same procedure will be performed while standing, by asking for strong straining and coughing, by increasing the intra-abdominal pressure, and visually visualizing whether there is urine leakage.
Urinary incontinence evaluated using the Uroflowmetry | change from baseline and 1, 2, and 3 months of practice
  The woman will be seated on the upper toilet, under which the uroflowmetric device is located, and the researcher will be asked to urinate completely with the "pee" command. After urinating completely, the process will be terminated with the "finish" command from the researcher. With this method, urination volume, flow duration, maximum flow rate, time to reach maximum speed, average flow rate and urination time values will be measured and the values will be taken through the software to which the device is connected.
Urinary incontinence evaluated using the Pelvic Floor Muscle Strength Measurement | change from baseline and 1, 2, and 3 months of practice
  With the device called "perinometry", which measures the pelvic floor muscle strength, the vaginal probe, which belongs only to the woman, will be placed 3 cm inside the chamber, and the pelvic floor muscle strength will be evaluated by giving the woman a muscle command to the pelvic floor muscles.
Urinary incontinence evaluated using the Digital Palpation | change from baseline and 1, 2, and 3 months of practice
  Digital Palpation is a subjective method applied by vaginal touch that evaluates the strength and endurance (maximum duration of contractions) of the pelvic floor muscles. Evaluation by digital palpation will be performed using the Modified Oxford Classification. Evaluation of PTK strength by digital examination (Modified Oxford scoring) PTK strength Muscle strength 0: No contraction Muscle strength 1: Contraction is minimal, able to hold fingers for less than 1 second. Muscle strength 2: Contraction is weak, there is no elevation of the fingers and can hold for 1-3 seconds. Muscle strength 3: With contraction, the doctor's fingers are lifted up to the posteriorvaginal wall, can hold for 4-6 seconds, can repeat 3 times. Muscle strength 4: The doctor's fingers rise up to the posterior vaginal wall, there is a feeling of more intense pressure on the fingers and can hold it for 7-9 seconds, repeating it 3 times. Muscle strength 5: Can make one strong contraction lasting 10 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No